CLINICAL TRIAL: NCT07398911
Title: 3-Dimensional Simulation Guided Transcatheter Aortic Valve Replacement in Aortic Regurgitation(DIGITAL)
Acronym: DIGITAL
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Fu Wai Hospital, Beijing, China (Other); West China Hospital (Other); Beijing Anzhen Hospital (Other); General Hospital of Ningxia Medical University (Other); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Henan Provincial Chest Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Fujian Medical University Union Hospital (Other); Guangdong Provincial People's Hospital (Other); Xinqiao Hospital of Chongqing (Other); The Affiliated Hospital of Qingdao University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Yan'an Hospital of Kunming City (Unknown); Dong'e People's Hospital (Unknown)
Responsible Party: Principal Investigator, Jian Yang, Chief Physician, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TAVR-AR-3D
Record Dates: First submitted 2025-04-10; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Aortic Regurgitation
Keywords: Aortic Regurgitation; transcatheter aortic valve replacement; 3D simulation technology; DIGITAL
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): Using 3D simulation technique
  Interventions: Device: 3D simulation technique
- Control group (No Intervention): Not using 3D simulation technique

INTERVENTIONS:
Device: 3D simulation technique — using 3D simulation technique
  Arms: Test group

SUMMARY:
This study will evaluate the safety and efficacy of postmarket bioprosthetic aortic valve in patients with severe aortic regurgitation undergoing transapical transcatheter aortic valve replacement based on 3D simulation technology using a prospective, randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* All of the following conditions must be met for inclusion:

  1. Age ≥ 65 years;
  2. Symptomatic severe native aortic regurgitation;
  3. Aortic valve anatomy assessed by investigator as suitable for transcatheter aortic valve replacement ;
  4. Subjects signed a written informed consent and agreed to cooperate with all follow-up examinations.

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria were not included:

  1. Active endocarditis;
  2. Acute myocardial infarction or unstable angina pectoris, or severe coronary stenosis requiring coronary revascularization within 3 months;
  3. Stroke or TIA (transient ischemic attack) within the past 3 months;
  4. Any intracardiac mass, left ventricular or atrial thrombus, vegetation detected by echocardiography;
  5. Severe obstructive hypertrophic cardiomyopathy (LVOTG peak ≥ 30 mmHg at rest); Note: Literature Basis: Chinese Guidelines for the Diagnosis and Treatment of Hypertrophic Cardiomyopathy 2023
  6. History of bleeding tendency or coagulopathy or refusal of blood transfusion;
  7. Active gastric ulcer or active gastrointestinal (GI) bleeding within 3 months;
  8. Presence of contraindication to anticoagulation or antiplatelet;
  9. Complicated with severe other valve diseases requiring concurrent surgical intervention;
  10. Prior aortic valve graft (mechanical or bioprosthetic);
  11. Severe left ventricular dysfunction, left ventricular ejection fraction < 30%;
  12. Hepatic encephalopathy or acute active hepatitis;
  13. Renal dysfunction (eGFR < 30ml/min calculated according to Cockcroft-Gault formula) and/or ongoing renal replacement therapy;
  14. Patients with severe dementia and other poor compliance, unable to ensure the completion of the investigator;
  15. Emergency surgery required for any reason;
  16. Known hypersensitivity to contrast agents or nitinol memory alloys or porcine products;
  17. Patients who are pregnant or plan to become pregnant, or are taking estrogen or estrogen-like drugs (women suspected of becoming pregnant must have a negative serum or urine test for human chorionic gonadotropin before being included in the study);
  18. Other patients considered unsuitable for this clinical study by the investigator;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 354 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Coaxial ratio of prosthetic aortic valve | 12 months
  Definition: A coaxial index of less than 4 degrees or a coaxial angle of less than 10 degrees is considered coaxial if one of them is met, and the ratio of coaxial prosthetic aortic valves in the two groups test group (with 3D simulation technique) or control group (without 3D simulation technique) is calculated, respectively Coaxial rate per group = number of coaxial aortic valve prostheses per group/total number of cases per group 100%

SECONDARY OUTCOMES:
All-cause death, Disabling stroke, Myocardial infarction, and Heart failure | 30 days
  Number of patients that had any of these events
Technical success | immediate postoperative
  No operative mortality;Successful puncture, device delivery and delivery system retrieval;Correct positioning and release of a single bioprosthetic aortic valve to the appropriate anatomical location;No device-related procedures or interventions, no major vascular or access-related complications, and no structural cardiac complications
All-cause mortality | 30 days,12 months
  Rate of all-cause mortality
Device success | 30 days
  Technical success • Freedom from death • No device-related procedures or interventions, no major vascular or access-related complications, and no structural cardiac complications • The performance of the bioprosthetic aortic valve meets clinical requirements (mean aortic valve gradient < 20 mmHg, peak velocity < 3 m/s, Doppler velocity index ≥0.25 and < moderate aortic regurgitation)
Myocardial infarction | before discharge, 30 days, 12 months
  Number of patients that had event
Incidence of coronary obstruction | before discharge
  Number of patients that had event
CT imaging changes | 12 months
  1) New aortic sinus volume formed after prosthetic valve implantation2) Low density leaflet thickening/leaflet thrombosis on prosthetic valve
New York Heart Association Functional Classification | before discharge, 30 days , 12 months
Evaluation cardiac function by electrocardiography | 30 days,12 months
  Left ventricular ejection fraction (%)
Evaluation cardiac function by electrocardiography | 30 days,12 months
  Left ventricular end diastolic diameter (mm)
Evaluation of bioprosthesis performance by echocardiography | 30 days,12 months
  Using the following measures:Aortic Valve Mean Gradient (cm2)
Evaluation of bioprosthesis performance by echocardiography | 30 days,12 months
  Using the following measures:Transaortic peak velocity
Evaluation of bioprosthesis performance by echocardiography | 30 days,12 months
  Using the following measures:Transaortic Central Regurgitation Severity
Evaluation of bioprosthesis performance by echocardiography | 30 days,12 months
  Using the following measures:Perivalvular Leak Severity
Contents of evaluation: including valve displacement, valve embolism and ectopic valve deployment | immediate postoperative
  Valve Dislodgement: Following initial correct positioning, the prosthesis moved upward or downward within the aortic annulus from its initial position without valve embolization Valve embolization: Prosthesis moves upward or downward after final deployment, thereby losing contact with the aortic annulus Ectopic Valve Deployment: Prosthesis deployed in unintended location and unable to be explanted due to valve embolization or inability to deliver valve to intended location
Major Cardiac Structural Complications | before discharge, 30 days
  Number of patients that had these events

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China